CLINICAL TRIAL: NCT02165761
Title: Evaluation of Anti-platelet Factor 4/Heparin Antibodies in Hemodialysis Patients Implanted With the GORE® Hybrid Vascular Graft Versus Non-heparin Bonded Synthetic Vascular Grafts.
Brief Title: Evaluation of Anti-platelet Factor 4/Heparin Antibodies in Hemodialysis Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HVG 13-01
Record Dates: First submitted 2014-06-13; First posted 2014-06-17 (Estimated); Results first posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: End Stage Renal Disease
Keywords: Hemodialysis; End Stage Renal Disease; Vascular Graft
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GORE® Hybrid Vascular Graft (Active Comparator): GORE® Hybrid Vascular Graft
  Interventions: Device: GORE® Hybrid Vascular Graft
- Non-heparin bonded synthetic graft (Other): Non-heparin bonded synthetic graft
  Interventions: Device: Non-heparin bonded synthetic graft

INTERVENTIONS:
Device: GORE® Hybrid Vascular Graft
  Arms: GORE® Hybrid Vascular Graft
Device: Non-heparin bonded synthetic graft
  Arms: Non-heparin bonded synthetic graft

SUMMARY:
To characterize the GORE® Hybrid Vascular Graft as compared to non-heparin bonded synthetic vascular grafts in terms of the prevalence and persistence of anti-platelet factor 4 / heparin antibodies (anti-PF4 / H antibodies).

ELIGIBILITY:
Inclusion Criteria:

* The patient is not a candidate for a native fistula.
* The patient requires the creation of an upper arm vascular access graft for hemodialysis secondary to a diagnosis of End-Stage Renal Disease.
* The patient has been on hemodialysis for ≥1 month.

Exclusion Criteria:

* The patient is scheduled for a different surgical procedure within 30 days post Index Procedure.
* The patient has a known hypercoagulable disorder or bleeding disorder.
* The patient has had a previous instance of Heparin Induced Thrombocytopenia Type II (HIT type II) or has known sensitivity to heparin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-07; Primary Completion 2017-01-20 (Actual); Study Completion 2017-01-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Hackensack, New Jersey
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- GORE® Hybrid Vascular Graft: Subjects Randomized to the GORE® Hybrid Vascular Graft
- Non-heparin Bonded Synthetic Graft: Subjects Randomized to the Non-heparin bonded synthetic graft
Period: Overall Study
Arm/Group | GORE® Hybrid Vascular Graft | Non-heparin Bonded Synthetic Graft
Started | 23 | 19
Completed | 4 | 5
Not Completed | 19 | 14

BASELINE CHARACTERISTICS:
Groups:
- GORE® Hybrid Vascular Graft: GORE® Hybrid Vascular Graft>
  > GORE® Hybrid Vascular Graft
- Non-heparin Bonded Synthetic Graft: Non-heparin bonded synthetic graft>
  > Non-heparin bonded synthetic graft
- Total: Total of all reporting groups
Arm/Group | GORE® Hybrid Vascular Graft | Non-heparin Bonded Synthetic Graft | Total
Number analyzed (Participants) | 23 | 19 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (12.9) | 58.7 (12.2) | 60.4 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 9 | 23
  Male | 9 | 10 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 23 | 19 | 42
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 15 | 34
  White | 4 | 4 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 19 | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Prevalence of a Positive Poly-specific Enzyme Immunoassay (EIA) at Day 7 and/or Day 14 Time Points
Description: Antibody screening was performed using a commercial poly-specific EIA that detects antibodies of any of the IgG, IgA, and / or IgM classes against PF4/polyvinyl sulfonate complexes, the EIA-GAM.
Time Frame: 14 days after index procedure
Population: In the GORE® Hybrid Vascular Graft Group 19 out of 23 participants had obtained a serology sample at Day 7 and/or Day 14 for analysis.
  In the Non-heparin bonded synthetic graft Group 16 out of 19 participants had obtained a serology sample at Day 7 and/or Day 14 for analysis.
Measure: Count of Participants; unit: Participants
Groups:
- GORE® Hybrid Vascular Graft: GORE® Hybrid Vascular Graft >
  > GORE® Hybrid Vascular Graft
- Non-heparin Bonded Synthetic Graft: Non-heparin bonded synthetic graft >
  > Non-heparin bonded synthetic graft
Arm/Group | GORE® Hybrid Vascular Graft | Non-heparin Bonded Synthetic Graft
Number analyzed (Participants) | 19 | 16
Participants | 3 | 2

ADVERSE EVENTS:
Time Frame: 2 years, 3 months
Groups:
- Hybrid Vascular Graft (Test): Hybrid Vascular Graft (Test)
- Non-Heparin Synthetic Graft (Control): Non-Heparin Synthetic Graft (Control)
Arm/Group | Hybrid Vascular Graft (Test) | Non-Heparin Synthetic Graft (Control)
All-Cause Mortality (participants affected / at risk) | 1/23 | 1/19
Serious Adverse Events (participants affected / at risk) | 6/23 | 5/19
Other Adverse Events (participants affected / at risk) | 4/23 | 8/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hybrid Vascular Graft (Test) (N=23) | Non-Heparin Synthetic Graft (Control) (N=19)
Unsteady gait (General disorders) | 1 | 0
Weakness (General disorders) | 1 | 0
Cellulitis of legs (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 1 | 0
Graft infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 0 | 1
Sigmoid diverticulitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Motor vehicle accident (Injury, poisoning and procedural complications) | 1 | 0
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 | 0
Adult failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion recurrent (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Hybrid Vascular Graft (Test) (N=23) | Non-Heparin Synthetic Graft (Control) (N=19)
Peripheral edema (General disorders) | 0 | 1
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 1 | 1
Venous pressure increased (Investigations) | 0 | 1
Numbness in hand (Nervous system disorders) | 0 | 1
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Hematoma (Vascular disorders) | 0 | 1
Steal syndrome (Vascular disorders) | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Statistical Analysis Plan (2015-02-21): https://cdn.clinicaltrials.gov/large-docs/61/NCT02165761/SAP_000.pdf
  • Study Protocol (2014-11-06): https://cdn.clinicaltrials.gov/large-docs/61/NCT02165761/Prot_001.pdf